CLINICAL TRIAL: NCT05081375
Title: A Blinded, Controlled, Randomized Study of the Safety of Pre-operative Enoxaparin in the Surgical Management of Multi-trauma Patients Undergoing Orthopedic Surgical Procedures
Brief Title: Pre-operative Enoxaparin in the Surgical Management of Multi-trauma Patients Undergoing Orthopedic Surgical Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Valleywise Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-071
Record Dates: First submitted 2020-01-16; First posted 2021-10-18 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Venous Thrombosis Deep (Limbs); Surgical Blood Loss
Keywords: prophylaxis of DVT
MeSH Terms: conditions — Venous Thrombosis; Blood Loss, Surgical | interventions — Enoxaparin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Blinded, Controlled, Randomized, Safety Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding will be done by research pharmacist. Nurse Manager will also be un-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enoxaparin (Active Comparator): Enoxaparin dose will not be held for surgical procedure.
  Interventions: Drug: Enoxaparin Injectable Product
- Placebo dose given and Enoxaparin dose held (Placebo Comparator): Enoxaparin dose will be held and replaced by placebo and not given prior to surgical procedure.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Enoxaparin Injectable Product — Not holding prophylaxis dose prior to surgical procedure
  Other Names: Lovenox
  Arms: Enoxaparin
Drug: Sodium chloride — Holding prophylaxis dose of Enoxaparin replacing with placebo
  Other Names: Placebo
  Arms: Placebo dose given and Enoxaparin dose held

SUMMARY:
All trauma patients receive Lovenox or other prophylactic medication to prevent deep vein clots from forming. For the trauma patients with orthopedic injuries requiring surgery there is controversy over safety and efficacy when prophylaxis is started preoperatively vs postoperatively. This study is to evaluate both approaches for safety in terms of bleeding events during and 24 hours after surgery as well as preventing deep vein clot formation. This will be a randomized double blinded study using Lovenox or placebo as the medications given preoperatively. Postoperative Lovenox will be given to both groups per routine regime.

DETAILED DESCRIPTION:
This study will be conducted in an Intensive Care Unit (ICU) and Operating Room (OR) of Valleywise Health Medical Center. The study population will include adult subjects age ≥ 18 years of age, that require surgery for management of their traumatic long bone and/or pelvic fractures.

A total of 60 evaluable subjects will be enrolled in this pilot safety study, with a 1:1 randomization into each group. It is anticipated that approximately 70 patients will need to be consented to reach 60 evaluable subjects.

Subjects recruited for study participation must meet all study enrollment criteria prior to being enrolled in the study. Patients who meet inclusion / exclusion criteria will be invited to participate in the study. As feasible, the patient or his/her representative will be approached for enrollment in the study and asked to provide informed consent for participation.

Written informed consent will be obtained for all subjects by an investigator or delegate prior to enrollment in the study. All subjects meeting inclusion/exclusion criteria will be randomized to either enoxaparin or placebo.

Patients will be monitored for bleeding complications from the time of test article administration to 24 hours post-surgery. Subjects will be monitored for the development of DVT and/or PE through-out their hospitalization.

Subjects will be randomized to either 30 mg enoxaparin Sub Cutaneous (SQ) of 0.9% Sodium Chloride (NaCl) placebo SQ. Randomization will be 1:1, using a masked randomization list. Study personnel and the treatment team will be blinded to the randomization assignment. The Clinical Research Manager and pharmacy staff will be un-blinded and will not participate in study assessments.

The two groups will be treated as follows:

Treatment Group:

Enoxaparin 30mg/0.3ml SQ will be given within 12 hours prior to surgery. If surgery should be delayed longer than 12 hours following the initial dose a second dose will be given to ensure uninterrupted dosing.

If the patient is already on Lovenox 12 hours prior to surgery, no doses will be skipped.

Placebo Group Normal Saline (0.9%) 0.3 ml SQ will be given within 12 hours prior to surgery If surgery should be delayed longer than 12 hours following the initial dose a second dose of normal saline will be given to ensure the appearance of uninterrupted dosing in order to maintain the blind.

If the patient is already being given Enoxaparin 12 hours prior to surgery, the dose 12 hours prior to surgery will be substituted with normal saline.

Both groups

Will receive routine administration of Enoxaparin 12 hours following surgery

Will be monitored at 12 hours and 24 hours post procedure for any evidence of deep vein thrombosis (DVT) or pulmonary embolism (PE) formation.

Will be monitored during surgery, at 12 hrs and 24 hrs post-operatively for any bleeding events. A bleeding event is present if one or more of the following are present:

A drop of 3mg/dl or more in hemoglobin, Transfusion of blood product, Intervention/surgery for bleeding (hematoma, hemorrhage)

The following information will be collected and recorded:

Demographics: name, age, race, ethnicity, height, weight, physical exam

1. Medical history
2. Acute trauma history
3. Surgical data: procedure, length of surgery, estimated blood loss
4. Lab results
5. Imaging results
6. Bleeding complications
7. DVT and PE events
8. Outcome data (length of stay, ICU days, vent days, complications, disposition, etc.)
9. Unanticipated problems

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Traumatic injury of long bones or pelvis requiring surgical intervention
* Admission to the ICU

Exclusion Criteria:

* Age < 18 years
* Intracranial hemorrhage
* Direct admit to OR without prior ICU admission
* Pregnancy
* Prisoner
* Chronic Kidney Disease requiring dialysis or a glomerular filtration rate (GFR) or creatinine clearance requiring a decrease in Enoxaparin dosage
* Presence of DVT prior to study drug dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Evaluate Bleeding Complications Related to DVT chemoprophylaxis | From the time of study drug administration to 24 hours post-operation
  Evaluate the rate of bleeding complications related to DVT chemoprophylaxis after administering DVT chemoprophylaxis vs holding doses within 12 hours of surgery in patients with long bones and/or pelvic fractures requiring surgical intervention.
Evaluate Other Complications (besides bleeding) Related to DVT chemoprophylaxis | From the time of study drug administration to 24 hours post-operation
  Evaluate the rate of other complications (besides bleeding) Related to DVT chemoprophylaxis after administering DVT chemoprophylaxis vs holding doses within 12 hours of surgery in patients with long bones and/or pelvic fractures requiring surgical intervention.

SECONDARY OUTCOMES:
Incidence of DVT and PE | From the time of study drug administration to hospital discharge up to 3 months
  Recording any incidence of deep vein thrombosis or pulmonary embolism
study duration | From Institutional Review Board approval to date of last subject completion up to 2 years
  Record the time required to complete study enrollment goals
Assess feasibility of a larger trial with respect to study design | Duration of the study up to 2 years
  Assess a superiority study design using the rates of development of DVT/PE.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wertin, MD, FACS, Principal Investigator — Valleywise Health
Locations (1):
- Valleywise Health, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No